CLINICAL TRIAL: NCT07357363
Title: REThink for Mental Health of the Youths in Romania
Brief Title: REThink for Mental Health of Youths in Romania
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Oana David, Professor Ph.D of Clinical Psychology, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REThinkBullying Being
Record Dates: First submitted 2026-01-15; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Bullying Victimisation; Bullying of Child; Bullying Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: REThink (Experimental): To ensure age-appropriate interventions, students below the age of 18 in the experimental group will receive the REThink game, while college-aged participants will engage with the REThink LIFE game.
  Interventions: Behavioral: REThink Intervention
- Control (No Intervention): The students randomized in the control group will access the intervention after finalizing the post-test measurement

INTERVENTIONS:
Behavioral: REThink Intervention — At its core, the REThink game consists of seven levels, each focusing on a specific emotion-regulation skill crucial for emotional health. The game's story is based on the RETMAN character which helps the player fight the power of the "Irrationalizer" who personalizes irrational beliefs. The game is based on cognitive-behavioral psychotherapy - the unified protocol (Barlow et al., 2004) and well-supported Rational Emotive Behavioral Therapy (Ellis, 1995). Each level is composed of three sublevels, increasing in difficulty, and also has an embedded validated assessment system (composed of a sublevel for each level; David, Tomoiaga & Fodor, 2024), and can function as a standalone intervention.
  Arms: Experimental: REThink

SUMMARY:
In order to test the effect of the intervention, a multi-center randomized control trial (RCT) will be conducted to test the efficacy of the REThink interventions on improving bullying (both victimization and aggression) and mental health compared with a care as usual group. A minimum of 1000 students from the participating institutions (schools will be able to join based on a recruitment call), will be recruited and randomly assigned to either the experimental or control group.

ELIGIBILITY:
Inclusion Criteria:

* internet and PC access to complete the scales and game

Exclusion Criteria:

* no internet of PC access

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Bullying | baseline assessment, one week before starting the intervention
  Bullying and Cyberbullying Scale for Adolescents will be used to measure bullying. The scale is composed of 26 items, the minimum score is 26 and the maximum 130. Higher scores represent higher levels of bullying
Mental Health | baseline assessment
  Depression, Anxiety, and Stress Scale is used for mental healh. For this scale, lower scores represent lower levels of anxiety, depression and stress, the minimum score is 0 and maximum score is 63.
Mental Health Stigma | baseline assessment
  Peer Mental Health Stigmatization Scale measures mental health stigma. Lower scores represent an improvement.
Stress | baseline assessment
  MoodWheel instrument is used to measure stress. The scale is composed of 32 items representing emotions which are divided into four subscales: positive functional emotions, positive dysfunctional emotions, negative functional and negative dysfunctional emotions. Scores at each subscale represent higher levels of that category of emotion.The minimum score is 0 and the maximum is 160.
Self Compassion | baseline assessment
  The Self-Compassion Scale Short Form is used to measure self-compassion. The scale has two dimensions, namely Self-Care, where higher scores represent higher levels of self-care, and Self-Disparagement, where lower scores represent an improvement.The minim score is 12 and the maximum is 60.
Compassion | baseline assessment, one week before starting the intervention
  Compassion Scale for children is a valid and reliable measurement tool that will be able to determine the level of compassion of children between the ages of 10 to 18-year-olds.The minimum score is 9, and maximum is 54.
Emotion Regulation | baseline assessment, one week before starting the intervention
  The in-game assessment for each REThink intervention. This assessment system is the trial version of the game with sections for each level and very good psychometric properties. For this system, higher scores represent higher levels of various emotion-regulation abilities.
Trauma Screening | baseline assessment, one week before starting the intervention
  Childhood Trauma Screener is used to measure past traumatic experiences .The scale is composed of 5 items each representing a type of trauma or abuse. Higher scores represent higher frequency of abuse and/or trauma. The minimum score is and the maximum score is 5 and the maximum 25.
Changes in Bullying | post-test assessment, one week after finishing the intervention
  Bullying and Cyberbullying Scale for Adolescents will be used to measure bullying. The scale is composed of 26 items, the minimum score is 26 and the maximum 130. Higher scores represent higher levels of bullying
Changes in Mental Health | post-test assessment, one week after finishing the intervention
  Depression, Anxiety, and Stress Scale is used for mental healh. For this scale, lower scores represent lower levels of anxiety, depression and stress, the minimum score is 0 and maximum score is 63.
Changes in Mental Health Stigma | post-test assessment, one week after finishing the intervention
  The Peer Mental Health Stigmatization Scale measures mental health stigma. Lower scores represent an improvement.
Changes in Stress | post-test assessment, one week after finishing the intervention
  MoodWheel instrumentis used to measure stress. The scale is composed of 32 items representing emotions which are divided into four subscales: positive functional emotions, positive dysfunctional emotions, negative functional and negative dysfunctional emotions. Scores at each subscale represent higher levels of that category of emotion.The minimum score is 0 and the maximum is 160
Changes in Self-Compassion | post-test assessment, one week after finishing the intervention
  The Self-Compassion Scale Short Form is used to measure self-compassion. The scale has two dimensions, namely Self-Care, where higher scores represent higher levels of self-care, and Self-Disparagement, where lower scores represent an improvement.The minim score is 12 and the maximum is 60.
Changes in Compassion | post-test assessment, one week after finishing the intervention
  Compassion Scale for children is a valid and reliable measurement tool that will be able to determine the level of compassion of children between the ages of 10 to 18-year-olds.The minimum score is 9, and maximum is 54.
Changes in Emotion Regulation | post-test assessment, one week after finishing the intervention
  The in-game assessment for each REThink intervention. This assessment system is the trial version of the game with sections for each level and very good psychometric properties. For this system, higher scores represent higher levels of various emotion-regulation abilities.

CONTACTS AND LOCATIONS:
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: Undecided